CLINICAL TRIAL: NCT07193173
Title: Is the Two-minute Step Test an Alternative to the Six-minute Walk Test in Pulmonary Hypertension?: Validation of 2 Minute Step Test
Brief Title: Is the Two-minute Step Test an Alternative to the Six-minute Walk Test in Pulmonary Hypertension?
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Pinar BASTURK MERC, Principal Investigator, Physiotherapist, PhD, Saglik Bilimleri Universitesi
Other Study IDs: 2460
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; 2 minute step test; 6 minute walk test; validation
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 2 minute step test — The 2-Minute Step Test (2MST) is a simple, validated field test used to assess aerobic endurance and functional fitness, especially in older adults or people with chronic conditions (e.g., cardiopulmonary disease, neurological disorders).

SUMMARY:
The aim of this observational study is to evaluate the validity of the 2-minute step test in assessing functional capacity in pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a progressive cardiopulmonary disorder characterized by elevated pulmonary artery pressure, which can lead to right ventricular dysfunction and ultimately heart failure. Right heart catheterization is used to diagnose the disease, and individuals are diagnosed with PH when the mean pulmonary artery pressure is 20 mmHg or higher. Exercise intolerance is one of the key features of PH. The 6-minute walk test (6MWT) is the most commonly used test method in PH centers for assessing functional exercise capacity and plays a key role in the evaluation and management of PH. However, it has significant limitations in this context. Although the 6MWT is currently recommended for assessing functional exercise capacity independently of the environment, it is not feasible in most clinics, homes, and medical offices due to the requirement for a 30-meter-long corridor. The long-standing need for a practical and effective exercise assessment tool that is independent of physical space highlights the need for new methods to assess functional capacity. The 2-minute walk test was developed by Rikli and Jones in 1999.

The test requires individuals to stand and step in place as quickly as possible for 2 minutes while raising their knees to a height between the patella and iliac crest. Performance in the test is defined as the number of steps taken on the right side within 2 minutes, reaching the criterion height. The validity and reliability of the 2-minute step test have previously been investigated in patients with back pain, cardiopulmonary rehabilitation patients, and hypertensive geriatric patients.

The aim of this study is to evaluate the validity of the 2-minute step test in assessing functional capacity in PH.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with pulmonary hypertension (PH)
* Being 18 years of age or older
* Agreeing to participate in the study

Exclusion Criteria:

* Acute decompensated heart failure
* Orthopedic or neurological disorders that prevent the test from being performed
* Patients who have difficulty understanding the instructions given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being diagnosed with pulmonary hypertension (PH)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
2 Minute Step Test | 2 minutes
  The 2-minute step test (2MST) is a test used to assess functional capacity. The maximum number of knee lifts the individual can perform within 2 minutes will be counted, with the minimum height occurring at the midpoint between the patella and the anterior superior iliac spine (during steady walking, without changing position). The test will be performed with a mobile ergospirometer (K5, Cosmed, Italy). Oxygen consumption, task-based heart rate, and ventilation obtained during the 2MST will be recorded. In addition, the Borg dyspnea and fatigue scale will also be included in the assessment.

SECONDARY OUTCOMES:
Functional capacity | 6 minutes
  The 6-minute walk test will be performed.
mMRC Dyspnea Scale | 5 minutes
  This scale is a five-item scale (0: no dyspnea, 4 severe dyspnea) based on various physical activities that cause the feeling of dyspnea. Here, patients are asked to mark the level of activity that causes dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The sharing of this information is restricted by the ethics committee and informed consent form.